CLINICAL TRIAL: NCT00029185
Title: Topical Dehydrex in Treating Recurrent Corneal Erosion
Brief Title: Study of Dehydrex in Patients With Corneal Erosion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Holles Laboratories, Inc. (Industry)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: FD-R-1984-01; FD-R-001984-01
Record Dates: First submitted 2002-01-08; First posted 2002-01-09 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2001-10

CONDITIONS: Corneal Diseases; Recurrence
Keywords: Corneal Erosion; Dextrans; Administration, Topical; Ophthalmic Solutions; Thimerosal
MeSH Terms: conditions — Corneal Diseases; Recurrence

INTERVENTIONS:
Drug: Dehydrex

SUMMARY:
This is a compassionate-use treatment study to provide Dehydrex to patients with corneal erosion syndrome who have previously used Dehydrex.

DETAILED DESCRIPTION:
This study continues to provide Dehydrex to patients who have received it previously under other studies. Patients continue to be treated with their current dose of Dehydrex. Upward dose adjustments may be made as clinically indicated. Patients undergo eye exams every 3 to 4 months or more often. Downward dose titration will be attempted in patients who are stable, free of symptoms, and willing to attempt downward adjustments. In patients who are able to discontinue the medication, duration of healing will be determined. In those patients who experience a recurrence after discontinuing the medication, Dehydrex will be restarted at a dose higher than the minimum effective dose. After at least 8 weeks of treatment and resolution of symptoms, the dose may again be reduced. Further attempts to discontinue the medication will not be made.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of symptomatic recurrent corneal syndrome due to anterior membrane dystrophy or posttraumatic abrasion
* Not responsive to standard medical therapy with artificial tears, hypertonic saline, or bandage soft contact lenses
* At least 3 episodes of erosion within the past 4 months documented by slit lamp examination

Exclusion criteria:

* Allergy to any component of the medications to be used
* Active ocular surface infection due to bacteria, virus, or fungus
* Chronic atopic disease affecting the ocular surface or adnexa
* Dry eye, exposure, trichiasis, entropion, ectropion, or neurotrophic keratopathy
* Concurrent use of contact lenses
* Diagnosis of persistent epithelial defect in eye to be treated
* Concurrent use of topical medication to eye to be treated
* Any ocular eyelid surgery within the past 6 months
* Pre-existing corneal stromal edema
* Diabetes mellitus
* Postsurgical infection
* Dry eye condition of 16 or greater on Patient's Dry Eye Questionnaire
* Other investigational medications within the past 6 months
* Other corneal dystrophy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2001-09; Study Completion 2007-09

CONTACTS AND LOCATIONS:
Locations (1):
- Holles Laboratories, Inc., Cohasset, Massachusetts, United States